CLINICAL TRIAL: NCT00283166
Title: Coaching to Improve Care of Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Kaiser Permanente (Other); VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 224690; RSGPB-06-091-01-CPPB; ACS-KRPC-0609 (Other: UC Davis)
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: Palliative Care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Tailored Coaching and Education
  Interventions: Behavioral: Tailored Education and Coaching
- B (Other): Active Control
  Interventions: Behavioral: Tailored Education and Coaching

INTERVENTIONS:
Behavioral: Tailored Education and Coaching — A: Patients receive one-on-one counseling and education about pain management and improving doctor-patient communication B: Patients receive booklet on cancer pain control

SUMMARY:
An estimate of 90% of patients with cancer experience at least moderate pain at some point in their illness, and 42% of patients do not receive adequate palliation. The main objective of this research is to reduce barriers to pain control by creating more effective partnerships between patients and their health care providers. The aims of the study are: 1) to compare the effects on pain, cancer-related symptoms, and health-related quality of life of a standard cancer pain leaflet versus face-to-face, tailored education and coaching; 2) to estimate the effect of tailored education and coaching on patients' self confidence for managing their pain and participating actively in care; and 3) to examine the mechanisms underlying the beneficial effects of the intervention. The proposed model will enhance research on pain management in that it is a pilot-tested intervention that is applicable in the outpatient setting, based on Social Cognitive Theory, and focused on patient activation and education.

DETAILED DESCRIPTION:
Background: A small, randomized trial was conducted in 2001, that supplied preliminary evidence that a carefully structured, one-time individualized education and coaching intervention has the potential to provide important clinical benefits for patients suffering from cancer-related pain. The study did not explore the impact of the intervention in a larger, more diverse patient population; the duration of the intervention's benefits; or the pathway by which the benefits are achieved. This project will attempt to address these issues while building on the literature that exists in palliation and physician-patient communication.

Objective/Hypothesis: The main objective of this research is to reduce barriers to pain control by creating more effective partnerships between patients and their health care providers.

Specific Aims: The aims of this study are: 1) to compare the effects on pain, cancer-related symptoms, and health-related quality of life of a standard educational intervention versus face-to-face, tailored education and coaching; 2) to estimate the effect of tailored education and coaching on self-efficacy for pain self-management and for participation in care; and 3) to examine the mechanisms underlying the beneficial effects of the intervention.

Study Design: The proposed study is a randomized, controlled trial comparing "education only" with tailored education and coaching for patient activation (TEC). Eligible patients scheduled to see their oncologist at any of the three participating health systems will be invited to participate in the study. Consenting patients will be randomly allocated to TEC or education only. The intervention will be applied during a brief session just before the scheduled oncology visit. Allocation will be concealed from physicians, interviewers, and data analysts. Patients assigned to the usual care group will review the content of a standard informational booklet on cancer pain. A health educator will review key learning points and be available to answer questions. Patients assigned to the TEC group will receive an intervention designed to improve self-efficacy for both pain self-management and participation in care. Data will be collected from patients in a private waiting alcove just prior to the index visit (personal interview); during the index visit (audio-taping); and then two, six, and 12 weeks after the visit (phone interview). In addition to assessing effectiveness of the intervention, the study is designed to measure potential mediators and intermediate outcomes (attitudes, beliefs, self-efficacy, patient participation, quality of care, and adherence) and to examine the mechanisms underlying the intervention's beneficial effects. The study will contribute to a test of Social Cognitive Theory by examining whether the benefit of the intervention is more powerfully attenuated by changes in attitudes and beliefs or by changes in self-efficacy.

Cancer Relevance: Uncontrolled cancer pain remains prevalent. An estimated 90% of patients with cancer experience at least moderate pain at some point in their illness, and 42% of patients do not receive adequate palliation. Aside from impairing quality of life, uncontrolled pain can contribute to depression, increase the likelihood of suicide, and decrease patient acceptance of potentially beneficial therapy. The proposed project is valuable in that it will confirm the benefit of patient coaching, elucidate its mechanisms, and test Social Cognitive Theory. The proposed model will enlarge existing research on pain management in that it is: a (1) pilot tested, easily implementable intervention that is (2) applicable in the outpatient setting, (3) based on strong theory that makes predictions about mechanisms of benefit, and (4) focused on patient activation as well as education.

ELIGIBILITY:
Inclusion Criteria:

* Seen or scheduled to be seen at participating facility
* Diagnosis of locally advanced or disseminated lung, breast, prostate, head and neck, gynecologic (ovarian, uterine, cervical), esophageal, or colorectal cancer
* English speaking
* Worst pain past two weeks 4/10 or higher

Exclusion Criteria:

* Major surgical procedure scheduled within six weeks
* Enrolled in hospice
* Followed by pain management service (more than one visit made or scheduled)
* Already contacted for study
* Positive six-item dementia screen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain control 2, 6, and 12 weeks after the index visit | Baseline, 2, 6, and 12 weeks

SECONDARY OUTCOMES:
Pain self-efficacy | Baseline, 2, 6, 12 weeks
Communication self-efficacy | Baseline, 2, 6, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Kravitz, MD, MSPH, Principal Investigator — UC Davis Center for Health Services Research in Primary Care
Locations (3):
- United States (3):
  - VA Northern California Health Care System, Mather, California
  - Kaiser Permanente Northern California, Oakland, California
  - UC Davis Cancer Center, Sacramento, California

REFERENCES:
- [Background] Kravitz RL, Tancredi DJ, Street RL Jr, Kalauokalani D, Grennan T, Wun T, Slee C, Evans Dean D, Lewis L, Saito N, Franks P. Cancer Health Empowerment for Living without Pain (Ca-HELP): study design and rationale for a tailored education and coaching intervention to enhance care of cancer-related pain. BMC Cancer. 2009 Sep 9;9:319. doi: 10.1186/1471-2407-9-319. PMID 19737424
- [Result] Street RL Jr, Slee C, Kalauokalani DK, Dean DE, Tancredi DJ, Kravitz RL. Improving physician-patient communication about cancer pain with a tailored education-coaching intervention. Patient Educ Couns. 2010 Jul;80(1):42-7. doi: 10.1016/j.pec.2009.10.009. Epub 2009 Dec 4. PMID 19962845